CLINICAL TRIAL: NCT02311517
Title: The Effects of Serratus Anterior Plane Block on Postoperative Quality of Recovery and Analgesia After Video-assisted Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2014-0853
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Quality of Recovery and Analgesia After Video-assisted Thoracoscopic Surgery
MeSH Terms: interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropivacaine group (Experimental): 45 patients will be randomly allocated into ropivacaine group with 0.4 ml/kg of 0.375% ropivacaine after induction of anesthesia.
  Interventions: Drug: Ropivacaine
- saline group (Placebo Comparator): 40 patients are randomly allocated into saline group with 0.4 ml/kg saline after induction of anesthesia.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Ropivacaine — 90 patients are randomly allocated into two groups: ropivacaine group (n=45), saline group (n=40). In the ropivacaine group, ultrasound-guided serratus anterior plane block is performed with 0.4 ml/kg of 0.375% ropivacaine after induction of anesthesia. In the saline group, ultrasound-guided serratus anterior plane block is performed with 0.4 ml/kg saline after induction of anesthesia.
  Arms: ropivacaine group
Drug: Normal Saline
  Arms: saline group

SUMMARY:
Postoperative pain still remains a challenging problem in patients undergoing video-assisted thoracoscopic surgery (VATS). However, there is no gold standard for regional analgesia for VATS. Serratus anterior plane block (SPB) under ultrasound guidance has been described recently to achieve complete paresthesia of the hemithorax. Therefore, SPB has the possibility to provide analgesia following thoracic surgery. Pain following surgery is a critical side effect of surgery, which increases the risk of complications and delays a recovery. Therefore, SPB may help not only reduce pain following VATS, but also increase the quality of recovery. This study aims to investigate the effectiveness of ultrasound-guided SPB on the quality of recovery and pain in patients undergoing VATS.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (20-65 years of age) scheduled for elective video-assisted thoracoscopic surgery
2. ASA class I and II

Exclusion Criteria:

1. Allergy to local anesthetics or contraindication to use of ropivacaine
2. Pregnancy
3. Neurologic and psychologic disease
4. Severe cardiovascular disease
5. Liver failure
6. Renal failure
7. Chronic treatment with analgesics

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-01-28; Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery 40 score | 24 hours after operation day

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea